CLINICAL TRIAL: NCT03076476
Title: Evaluation of Microcirculatory Protection In Percutaneous REvascularisation With Bioresorbable Vascular Scaffolds Versus Metallic Drug-eluting Stents: a Device- and Implant Technique-based Comparison
Brief Title: Coronary Microcirculatory and Bioresorbable Vascular Scaffolds
Acronym: EMPIRE-BVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P02135
Record Dates: First submitted 2017-01-26; First posted 2017-03-10 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: CHD - Coronary Heart Disease; Angina, Stable; Myocardial Ischemia
Keywords: Coronary Stent; PCI; BVS; Index of microcirculatory resistance
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Myocardial Ischemia | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DES-std group (Active Comparator): (DES: drug-eluting stent). Metallic DES implanted in standard fashion. To be compared with the DES-slow group at interim analysis at the end of phase 1 stage.
  Interventions: Device: Drug-Eluting Stent (DES) - standard(std)
- DES-slow group (Experimental): (DES: drug-eluting stent). Slow device inflation (mandated in the BVS IFU). To be compared with the DES-std group at interim analysis at the end of phase 1 stage.
  After the interim analysis DES-slow to be compared with BVS.
  Interventions: Device: Drug-Eluting Stent (DES) - slow
- BVS group (Experimental): (Bioresorbable Vascular Scaffold) Introduced after the interim analysis (phase 2) for comparison with DES-slow.
  Interventions: Device: Bioresorbable Vascular Scaffolds (BVS)

INTERVENTIONS:
Device: Bioresorbable Vascular Scaffolds (BVS) — Bioresorbable Vascular Scaffold. Introduced after the interim analysis (phase 2) for comparison with DES-slow.
  Other Names: ABSORB
  Arms: BVS group
Device: Drug-Eluting Stent (DES) - slow — Slow device inflation (mandated in the BVS IFU). To be compared with the DES-std group at interim analysis at the end of phase 1 stage.
  After the interim analysis DES-slow to be compared with BVS.
  Other Names: Xience
  Arms: DES-slow group
Device: Drug-Eluting Stent (DES) - standard(std) — Metallic DES implanted in standard fashion. To be compared with the DES-slow group at interim analysis at the end of phase 1 stage.
  Other Names: Xience
  Arms: DES-std group

SUMMARY:
Angina and heart attacks are caused by narrowings in the coronary arteries (blood vessels) supplying the heart. These narrowings can be opened using a balloon and stent (angioplasty). Traditionally, stents are constructed from metal and are permanent. However, newer stents are being constructed from carbohydrate polymers (scaffolds), which allow them to reabsorb over time leaving no permanent implant. New data has suggested that these scaffolds appear to reduce recurrent angina and may alter the blood flow down the artery. However, it is not known whether this is due to the scaffolds themselves or the way the scaffolds are inserted. In this study we hope to measure the blood flow to the heart and assess changes in that flow during stent and scaffold insertion. It is also important to know whether these effects are durable and thus, a cohort of patients will return at 3-months to be restudied. These data are important to help us understand why blood flow is affected by stent/scaffold selection or device implantation technique and whether this results in better long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age >18 years, <75 years.
2. Lesion suitability for BVS deployment: target vessel calibre >2.3mm and <3.8mm reference diameter, without significant tortuosity or calcification.
3. Listed for single-vessel PCI procedure.
4. Lesion length≤28mm (to accommodate single BVS/DES)
5. Preserved left ventricular ejection fraction (EF≥50%).

Exclusion Criteria:

1. Patients with confirmed myocardial infarction within the preceding 2 months.
2. Allergy or intolerance to aspirin, clopidogrel, prasugrel or ticagrelor or contraindication to 12 months' dual antiplatelet therapy.
3. Contraindication to use of adenosine (asthma/chronic lung disease with documented bronchoreactivity).
4. Significant known comorbidity or terminal condition with life expectancy <6 months.
5. Pregnancy.
6. Coagulopathy or warfarin treatment.
7. Significant renal impairment (baseline creatinine>130 mmol/l).
8. Other comorbid condition that may affect microcirculatory function or troponin release (eg. Seropositive inflammatory conditions).
9. Inability to comply with follow-up requirements.
10. Target lesion in left mainstem, saphenous vein or arterial grafts.
11. Chronic total occlusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Change in IMR between baseline and post-stent/scaffold implantation. | During procedure
  IMR: index of microvascular resistance
Change in CFR between baseline and post-stent/scaffold implantation. | During procedure
  CFR: coronary flow reserve

SECONDARY OUTCOMES:
Incidence of troponin elevation post-PCI (MI4a). | Measured 6 hours after stent insertion
  Measuring serum troponin I levels by blood test
Changes in IMR between baseline, post-implant and subsequent timepoints in subrandomized group. | 3 months follow up
  IMR: index of microvascular resistance
Incidence of post-PCI angina and quality of life by standardized Seattle angina questionnaire at telephone follow-up. | Up to 12 months
  Description: The Seattle Angina Questionnaire is a points based question and answer system where a overall score can be assessed and compared
Incidence of stent & scaffold expansion & malapposition adjudged by strut-level OCT analysis. | During index procedure and at 3 month follow up
  OCT analysis of stent struts done quantitatively
Incidence of stent/scaffold strut coverage/endothelialisation adjudged by strut-level OCT analysis. | During index procedure and at 3 month follow up
  OCT analysis of stent struts done quantitatively
Nature/phenotype of underlying target lesion plaque by OCT analysis. | During index procedure and at 3 month follow up
  OCT analysis of lesion characteristics done quantitatively
Adverse events | At time points 1, 3, 6 & 12 months post-PCI
  Adverse event assessed by clinical history and medical notes
Serious adverse events | At time points 1, 3, 6 & 12 months post-PCI
  Serious adverse event assessed by clinical history and medical notes

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Duckworth, Study Director — Papworth NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aetesam-Ur-Rahman M, Zhao TX, Paques K, Oliveira J, Chiu YD, Duckworth M, Khialani B, Kyranis S, Bennett MR, West NEJ, Hoole SP. Evaluation of microcirculatory protection in percutaneous revascularisation: A stent implantation technique and device comparison. Catheter Cardiovasc Interv. 2024 Sep;104(3):462-471. doi: 10.1002/ccd.31155. Epub 2024 Jul 24. PMID 39044651
- [Derived] Aetesam-Ur-Rahman M, Zhao TX, Paques K, Oliveira J, Khialani B, Kyranis S, Braganza DM, Clarke SC, Bennett MR, West NEJ, Hoole SP. Coronary Flow Variations Following Percutaneous Coronary Intervention Affect Diastolic Nonhyperemic Pressure Ratios More Than the Whole Cycle Ratios. J Am Heart Assoc. 2022 May 3;11(9):e023554. doi: 10.1161/JAHA.121.023554. Epub 2022 Apr 26. PMID 35470686